CLINICAL TRIAL: NCT00184366
Title: Classification and Characterization of Patients Suffering From Moderate to Severe Plaque Psoriasis Responding to Subcutaneous Administered Efalizumab
Brief Title: Classification and Characterization of Patients Treated With Efalizumab for Plaque Psoriasis
Status: Terminated | Type: Observational
Why Stopped: efalizumab was withdrawn from market; full 2 years follow-up only 14 patients
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: ROCAC
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Plaque Psoriasis
Keywords: drug therapy; efalizumab
MeSH Terms: interventions — efalizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: efalizumab — efalizumab

SUMMARY:
The main objectives of the project are:

* To classify patients suffering from plaque psoriasis responding on a given treatment (efalizumab) based upon reduction in Psoriasis Area and severity Index (PASI), Psoriasis Disability Index 8PDI) and dermatology Life Quality Index 8 DLQI)
* To characterize patients suffering from plaque psoriasis responding to or not responding to subcutaneous administrated efalizumab.

DETAILED DESCRIPTION:
This is an investigator initiated,prospective, longitudinal, observation study. Before starting treatment with efalizumab we will record factors such as demographic data, type of psoriasis, previous treatment, other diseases etc.

We will follow the patients and classify them as responders and non-responders. We hope to find 4-5 factors which we can use later to predict response of this drug.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe plaque psoriasis for more than six months
* eligible for efalizumab treatment according to current Norwegian guidelines

Exclusion Criteria:

* Pregnant or breast-feeding patients
* Patients with a history of uncontrolled bacterial, viral, fungal or atypical mycobacterial infection.
* Patients suffering from HIV, Hepatitis B or C, active tuberculosis, hepatic cirrhosis and hospital admission for cardiac disease, stroke or pulmonary disease within last year.
* Patients with history of cancer in the preceding 5 years, including lymphoproliferative disorders. patients with history of fully resolved basal cell or squamous cell skin cancer may be enrolled.
* Patients with impaired renal or hepatic function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of both genders, over the age of 18 years who have been suffering from moderate to severe plaque psoriasis for more than six months and who are eligible for efalizumab treatment according to current Norwegian guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2005-05; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Response PASI 75 | 2 years

SECONDARY OUTCOMES:
Dermatology Life Quality index (DLQI) | 2 years
Psoriasis disability Index (PDI) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Morten Dalaker, univ lekt II, Study Chair — St Olavs hospital, NTNU, Norway
Locations (1):
- Dep of dermatology, St Olavs Hospital, Trondheim, Norway